CLINICAL TRIAL: NCT05316948
Title: Mental Health and Sexuality in Adolescents and Young Adults
Acronym: SEX-T-ADO
Status: Recruiting | Type: Observational
Sponsor: Fondation Santé des Étudiants de France (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A03080-41
Record Dates: First submitted 2022-03-17; First posted 2022-04-07 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Psychiatric Disorder; Adolescent Behavior; Mental Health Issue
Keywords: psychotropic treatment; sexuality; teenagers and young adults
MeSH Terms: conditions — Mental Disorders; Adolescent Behavior; Sexuality

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: self-questionnaire — Quantitative survey with self-administered questionnaire offered to all patients attending psychiatry study care during the month of the assessment.

SUMMARY:
According to the World Health Organization (WHO), "Sexual health is a state of physical, emotional, mental and social well-being in relation to sexuality, not merely the absence of disease, dysfunction or of infirmity. Sexual health requires a positive and respectful approach to sexuality and sexual relationships [...]".

The main objective is to show that a training intervention intended for psychiatric care teams and targeted on the question of the impact of psychiatric disorders and psychotropic drugs on the sexuality of young people, increases the proportion of young people with whom the question of sexual health is discussed (in connection with psychiatric disorders and, if applicable, with the taking of psychotropic treatment, while they are hospitalized for a psychiatric disorder in the clinics of the FSEF and receive, or not, psychotropic treatment ).

DETAILED DESCRIPTION:
Non-interventional multicenter prospective mixed study (quantitative and qualitative).

Research process in 3 phases:

1. Inventory with a mixed method evaluation (quantitative survey and qualitative survey),

   * Step 1: quantitative survey with self-administered questionnaire offered to all patients attending psychiatric study care during the month of the assessment.
   * Step 2: qualitative survey of young people and caregivers.
2. Design and implementation of an intervention adapted to the needs of the field (training for caregivers and tools for young people).

   * Step 3: implementation of training programs for professionals based on data from phase 1 and preparation for interventions for young people.
   * Step 4: Interventions (interventions with young people in groups and individually).
3. Reassessment after the deployment of the intervention - Step 5: Finally, the quantitative survey of stage 1 with a self-questionnaire offered to all patients present in psychiatric care-study will be repeated during one month of the evaluation in order to measure the impact of the action taken.

ELIGIBILITY:
Inclusion Criteria:

* Young people hospitalized in psychiatric care-studies in one of the establishments of the FSEF,
* Age ≥ 15 years (age of sexual majority),
* Receiving or not a psychotropic treatment,
* No opposition to participation (or parents for minors) in the study and use of data

Exclusion Criteria:

* Refusal to participate
* Patient under 15 years old
* Need for emergency care (medicine or psychiatry).

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All young people hospitalized in the 13 structures of the FSEF aged 15 or over.
Sampling Method: Non-Probability Sample
Enrollment: 770 (Estimated)
Dates: Start 2023-02-27 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Comparison | self-questionnaire after the team training (T2 = 1 year)
  To show that a training intervention intended for the healthcare team makes it possible to increase the proportion of young people with whom the question of sexual health has been approached, in connection with psychiatric disorders and, if necessary, with taking treatment psychotropics; while they are hospitalized for a psychiatric disorder in the clinics of the FSEF and receive, or not, a psychotropic treatment.

SECONDARY OUTCOMES:
Description | self-questionnaire (T0 = within three months of the opening of the center)
  Describe the sexuality of adolescents and young adults hospitalized in a psychiatric establishment within the FSEF with quantitative survey with self-questionnaire exploring sexual adverse effects
Comparison | self-questionnaire (T0 = within three months of the opening of the center)
  To compare the sexual life of patients hospitalized at the FSEF for a psychiatric illness - according to whether or not they receive psychotropic treatment with quantitative survey with self-questionnaire exploring sexual adverse effects
Comparison | self-questionnaire after the team training (T2 = 1 year)
  To compare the perceived impact of psychiatric disorders and psychotropic treatments on patients' sexual satisfaction measured by a Likert scale of sexual satisfaction (rated from 1 to 5 with 1 equal to very satisfied and 5 to very dissatisfied) before and after intervention.

CONTACTS AND LOCATIONS:
Locations (12):
- France (12):
  - Clinique FSEF Vence, Vence, Alpes Maritimes
  - Clinique FSEF Grenoble La Tronche, Grenoble, Auvergne-Rhône-Alpes
  - Clinique FSEF Rennes-Beaulieu, Rennes, Brittany Region
  - Clinique FSEF Aire sur l'Adour, Aire-sur-l'Adour, Landes
  - Clinique FSEF Vitry-le-François, Vitry-le-François, Marne
  - Clinique FSEF Villeneuve d'Ascq, Villeneuve-d'Ascq, Nord
  - Clinique FSEF Sablé-sur-Sarthe, Sablé-sur-Sarthe, Pays de la Loire Region
  - Clinique FSEF Bouffémont, Bouffémont, Île-de-France Region
  - Clinique FSEF Neufmoutiers-en-Brie, Neufmoutiers-en-Brie, Île-de-France Region
  - Clinique FSEF Paris 13, Paris, Île-de-France Region
  - Clinique FSEF Paris 16, Paris, Île-de-France Region
  - Clinique FSEF Sceaux, Sceaux, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No